CLINICAL TRIAL: NCT02854566
Title: Periprosthetic Fractures of the Femur Treated by Osteosynthesis
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tamas Illes, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-Periprosthetic fractures
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Periprosthetic Fracture of the Femur
Keywords: periprosthetic fracture of the femur; hip prosthesis
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- periprosthetic fractures of the femur: periprosthetic fractures of the femur treated by osteosynthesis
  Interventions: Device: osteosynthesis

INTERVENTIONS:
Device: osteosynthesis — Fracture reduction and fixation with screws/plates/cables (standard of care)

SUMMARY:
Observational retrospective study on 36 consecutive patients having had surgery for a periprosthetic fracture of the femur between 2010 and 2015.

The goal of the study is to test whether osteosynthesis was a secure choice at a certain age and with any type of Vancouver fracture.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients having had surgery between 2010 and 2015 within the CHU Brugmann hospital for a periprosthetic fracture of the femur (osteosynthesis).

Exclusion Criteria:

* Death during surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Periprosthetic fractures of the femur treated by osteosynthesis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Age | Up to 2-3 days before surgery (pre-surgery radiography)
  Demographic data
Sex | Up to 2-3 days before surgery (pre-surgery radiography)
  Demographic data
Body Mass Index | Up to 2-3 days before surgery (pre-surgery radiography)
  Demographic data
Prosthesis type | Up to 2-3 days before surgery (pre-surgery radiography)
  PTH (total hip prosthesis) or BHP (bipolar hip prosthesis)
Type of fracture | Up to 2-3 days before surgery (pre-surgery radiography)
  Type of fracture according to the Vancouver International Classification
Femoral component | Up to 2-3 days before surgery (pre-surgery radiography)
  Need for cement within the femur or not
Time between 1st surgery and fracture | Up to 2-3 days before surgery (pre-surgery radiography)
  Time between 1st surgery and fracture
Fracture healing | 10 months after surgery
  Healing status of the fracture (healed/not healed)
Mortality rate | 10 months after surgery
  Mortality rate (any causes)
Complications rate | 10 months after surgery
  Total complications rate (local + systemic + implant)
ASA score | During surgery (up to 2 hours)
  ASA score
Blood loss | During surgery (up to 2 hours)
  Blood loss during surgery

SECONDARY OUTCOMES:
Laterality | Up to 2-3 days before surgery (pre-surgery radiography)
  Prosthesis on the right or on the left side

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Schiopu, MD, Principal Investigator — CHU Brugmann; Tamas Illes, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Gaski GE, Scully SP. In brief: classifications in brief: Vancouver classification of postoperative periprosthetic femur fractures. Clin Orthop Relat Res. 2011 May;469(5):1507-10. doi: 10.1007/s11999-010-1532-0. No abstract available. PMID 20809166
- [Background] Duncan CP, Haddad FS. The Unified Classification System (UCS): improving our understanding of periprosthetic fractures. Bone Joint J. 2014 Jun;96-B(6):713-6. doi: 10.1302/0301-620X.96B6.34040. PMID 24891568
- [Background] Lindahl H, Malchau H, Oden A, Garellick G. Risk factors for failure after treatment of a periprosthetic fracture of the femur. J Bone Joint Surg Br. 2006 Jan;88(1):26-30. doi: 10.1302/0301-620X.88B1.17029. PMID 16365115
- [Background] Laurer HL, Wutzler S, Possner S, Geiger EV, El Saman A, Marzi I, Frank J. Outcome after operative treatment of Vancouver type B1 and C periprosthetic femoral fractures: open reduction and internal fixation versus revision arthroplasty. Arch Orthop Trauma Surg. 2011 Jul;131(7):983-9. doi: 10.1007/s00402-011-1272-y. Epub 2011 Feb 18. PMID 21331551
- [Background] Learmonth ID. The management of periprosthetic fractures around the femoral stem. J Bone Joint Surg Br. 2004 Jan;86(1):13-9. No abstract available. PMID 14765858
- [Background] Corten K, Vanrykel F, Bellemans J, Frederix PR, Simon JP, Broos PL. An algorithm for the surgical treatment of periprosthetic fractures of the femur around a well-fixed femoral component. J Bone Joint Surg Br. 2009 Nov;91(11):1424-30. doi: 10.1302/0301-620X.91B11.22292. PMID 19880884
- [Background] Capello WN, D'Antonio JA, Naughton M. Periprosthetic fractures around a cementless hydroxyapatite-coated implant: a new fracture pattern is described. Clin Orthop Relat Res. 2014 Feb;472(2):604-10. doi: 10.1007/s11999-013-3137-x. PMID 23836241
- [Background] Niikura T, Sakurai A, Oe K, Shibanuma N, Tsunoda M, Maruo A, Shoda E, Lee SY, Sakai Y, Kurosaka M. Clinical and radiological results of locking plate fixation for periprosthetic femoral fractures around hip arthroplasties: a retrospective multi-center study. J Orthop Sci. 2014 Nov;19(6):984-90. doi: 10.1007/s00776-014-0622-3. Epub 2014 Aug 22. PMID 25145998
- [Background] Choo SK, Kim Y, Shin MJ, Oh HK. Conservative treatment after failure of internal fixation for periprosthetic femoral fractures: a report of two cases. Arch Orthop Trauma Surg. 2015 Jun;135(6):773-9. doi: 10.1007/s00402-015-2210-1. Epub 2015 Apr 18. PMID 25894000
- [Background] Baba T, Kaneko K, Shitoto K, Futamura K, Maruyama Y. Comparison of therapeutic outcomes of periprosthetic femoral fracture between treatments employing locking and conventional plates. Eur J Orthop Surg Traumatol. 2013 May;23(4):437-41. doi: 10.1007/s00590-012-1005-0. Epub 2012 May 17. PMID 23412148
- [Background] Muller FJ, Galler M, Fuchtmeier B. Clinical and radiological results of patients treated with orthogonal double plating for periprosthetic femoral fractures. Int Orthop. 2014 Dec;38(12):2469-72. doi: 10.1007/s00264-014-2464-1. Epub 2014 Aug 12. PMID 25109478
- [Background] Moloney GB, Westrick ER, Siska PA, Tarkin IS. Treatment of periprosthetic femur fractures around a well-fixed hip arthroplasty implant: span the whole bone. Arch Orthop Trauma Surg. 2014 Jan;134(1):9-14. doi: 10.1007/s00402-013-1883-6. Epub 2013 Nov 20. PMID 24253261